CLINICAL TRIAL: NCT06518941
Title: An Open Trial of a Novel Pharmacotherapy for Habit Modification in Anorexia Nervosa
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Joanna Steinglass, Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NKI2024-90
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa
Keywords: anorexia; anorexia nervosa; donepezil; eating disorders; acetylcholinesterase inhibitor; Acetylcholine; habit
MeSH Terms: conditions — Anorexia Nervosa; Anorexia; Feeding and Eating Disorders; Habits | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label (Experimental): Donepezil
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Study medication will be initiated at 1mg, to be taken before bed. Dosing will follow a flexible titration. The expected titration will be 1 mg for 2 weeks, 2.5 mg for 2 weeks, then 5 mg for 4 weeks. Doses may be lowered from those recommended by the protocol if side effects are significant.

SUMMARY:
The purpose of this study is to test the feasibility and tolerability of donepezil in a small group of patients with anorexia nervosa (AN). Study participants will be receiving care at the New York State Psychiatric Institute Eating Disorders Unit. Study medication will be increased from 1 mg per day to a maximum of 5 mg per day for up to 8 weeks. Participants will be closely monitored for side effects by a research psychiatrist every week, in addition to the regular clinical monitoring they receive during inpatient treatment. The study will also include assessments of habit strength to measure any changes in maladaptive eating habits over the course of the treatment.

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious mental illness affecting up to 4% of women in the United States, with a chronic course and a mortality rate 6 times that expected for young women (Arcelus et al., 2011). The core, salient behavior in AN is maladaptive food restriction that persists even after full weight restoration treatment (Steinglass et al., 2023). Pharmacologic approaches to the treatment of AN, to date, have attempted to capitalize on side effect profiles (e.g., weight gain) or efficacy in related disorders (e.g., depression) but have yielded disappointing results (Muratore and Attia, 2022). This program of research leverages advances in mechanism research, which has identified the importance of habit systems in AN (Conceição et al., 2023), to test whether a medication can target habitual restrictive intake and thereby help patients with AN.

Donepezil is an acetylcholinesterase inhibitor and an FDA-approved medication that has been shown to reverse habitual behaviors like excessive exercise and food restriction in a rodent model of AN. Donepezil has been studied for its potential effect in mitigating compulsive, habit-like symptoms in other clinical populations, with no adverse events (Bergman et al., 2016; Cubo et al., 2008). These data suggest that donepezil may be effective in reducing maladaptive behaviors in compulsive disorders. There is no control product in this study.

Study medication will be initiated at 1mg, to be taken before bed. Dosing will follow a flexible titration. The expected titration will be 1 mg for 2 weeks, 2.5 mg for 2 weeks, then 5 mg for 4 weeks. The target dose of 5 mg/day is lower than the approved dose for dementia and the dose used in a study of adults with Obsessive Compulsive Disorder (OCD) (Bergman et al., 2016). Doses may be lowered from those recommended by the protocol if side effects are significant.

The primary objective of this study is to test the feasibility and tolerability of donepezil among patients with AN. The exploratory objectives are to test the utility of donepezil to modify the habitual behaviors characteristic of AN.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study (Clinical interview).
3. Aged 18-60 years (Clinical interview).
4. Diagnosed with anorexia nervosa (EDA-5).
5. BMI ≥ 15 kg/m2 (Clinical team medical record)

Exclusion Criteria:

1. Score of High Risk on the Columbia Suicide Severity Scale (C-SSRS).
2. Pregnancy (Serum pregnancy test on admission).
3. Current diagnosis of schizophrenia, schizophreniform disorder, bipolar (type I), or substance use disorder (SCID).
4. Bradycardia (below 60 bpm) (vital signs measurement by the clinical team)
5. Corrected QT interval (QTc) greater than 480 ms at baseline (EKG).
6. Antipsychotic medication (antidepressants at a stable dose are allowed) (clinical interview).
7. Known allergic reactions to components of the donepezil (e.g., known hypersensitivity to donepezil hydrochloride) (clinical interview).
8. History of peptic ulcer disease (clinical interview).
9. History of arrhythmia (clinical interview).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Side Effects Form | From enrollment to the end of treatment at 8 weeks
  The study psychiatrist will assess the tolerability of donepezil during weekly meetings with participants. The presence of side effects will be assessed using the Side Effects Form. Higher scores indicate more severe side effects (each side effect is scored separately). The Clinical Global Impressions (CGI) scale will evaluate overall functioning and psychopathology.
Clinical Global Impressions Scale | From enrollment to the end of treatment at 8 weeks
  The Clinical Global Impressions Scale (CGI) is a seven-point scale. A score of 1 indicates the most positive change in the treatment course and the least severity of psychopathology, while a score of 7 indicates the most negative change in the treatment course and the highest severity of psychopathology.

SECONDARY OUTCOMES:
Self-Report Habit Index | From enrollment to the end of treatment at 8 weeks
  The Self-Report Habit Index (SRHI) is a 12-item scale that measures habit strength. Higher scores indicate greater habit strength.
Food Choice Task | From enrollment to the end of treatment at 8 weeks
  The Food Choice task is a computer based assessment of preferences for different foods. Higher scores indicate greater preferences. .

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study aims to include a small number of participants, and privacy and confidentiality will need to be considered against the benefits of data sharing.

REFERENCES:
- [Background] Attia E, Kaplan AS, Walsh BT, Gershkovich M, Yilmaz Z, Musante D, Wang Y. Olanzapine versus placebo for out-patients with anorexia nervosa. Psychol Med. 2011 Oct;41(10):2177-82. doi: 10.1017/S0033291711000390. Epub 2011 Mar 22. PMID 21426603
- [Background] Conceicao ISR, Garcia-Burgos D, de Macedo PFC, Nepomuceno CMM, Pereira EM, Cunha CM, Ribeiro CDF, de Santana MLP. Habits and Persistent Food Restriction in Patients with Anorexia Nervosa: A Scoping Review. Behav Sci (Basel). 2023 Oct 25;13(11):883. doi: 10.3390/bs13110883. PMID 37998630
- [Background] Cubo E, Fernandez Jaen A, Moreno C, Anaya B, Gonzalez M, Kompoliti K. Donepezil use in children and adolescents with tics and attention-deficit/hyperactivity disorder: an 18-week, single-center, dose-escalating, prospective, open-label study. Clin Ther. 2008 Jan;30(1):182-9. doi: 10.1016/j.clinthera.2008.01.010. PMID 18343255
- [Background] Steinglass JE, Fei W, Foerde K, Touzeau C, Ruggiero J, Lloyd C, Attia E, Wang Y, Walsh BT. Change in food choice during acute treatment and the effect on longer-term outcome in patients with anorexia nervosa. Psychol Med. 2024 Apr;54(6):1133-1141. doi: 10.1017/S0033291723002933. Epub 2023 Oct 2. PMID 37781904
- [Background] undefined
- [Background] El Mestikawy S, Wallen-Mackenzie A, Fortin GM, Descarries L, Trudeau LE. From glutamate co-release to vesicular synergy: vesicular glutamate transporters. Nat Rev Neurosci. 2011 Apr;12(4):204-16. doi: 10.1038/nrn2969. PMID 21415847
- [Background] Bergman J, Miodownik C, Lerner PP, Miodownik E, Shulkin A, Lerner V. Donepezil as Add-on Treatment for Resistant Obsessive-Compulsive Disorder: Retrospective Case Series. Clin Neuropharmacol. 2016 Jul-Aug;39(4):194-6. doi: 10.1097/WNF.0000000000000160. PMID 27223667
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255